CLINICAL TRIAL: NCT04416334
Title: PREEMPTIVE THERAPY WITH COLCHICINE IN PATIENTS OLDER THAN 60 YEARS WITH HIGH RISK OF SEVERE PNEUMONIAE DUE TO CORONAVIRUS SARS-CoV2 (COVID-19)
Brief Title: PREEMPTIVE THERAPY WITH COLCHICINE IN PATIENTS OLDER THAN 60 YEARS WITH HIGH RISK OF SEVERE PNEUMONIAE DUE TO CORONAVIRUS
Acronym: COLCHI-COVID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Collaborators: Gerencia de atención primaria área 1 (Unknown); Gerencia de atención primaria área 2 (Unknown); Gerencia Atencion Primaria Area 3 (Other Government); Gerencia de atención primaria área 4 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COLCHICOVID
Record Dates: First submitted 2020-06-03; First posted 2020-06-04 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: SARS-CoV-2 Infection (COVID-19)
Keywords: colchicine
MeSH Terms: conditions — COVID-19 | interventions — Colchicine; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine plus symptomatic treatment (paracetamol). (Experimental): Patients in this arm will receive study medication colchicines 0.5 mg orally (PO) twice daily for the first 3 days and then once daily for the last 18 days. If a dose is missed, it should not be replaced.
  All patients should also receive best symptomatic treatment (mainly paracetamol), based on clinical practice.
  Interventions: Drug: Colchicine plus symptomatic treatment (paracetamol)
- Symptomatic treatment (Active Comparator): Symptomatic treatment (paracetamol or best symptomatic treatment based on doctor recommendations).
  Interventions: Drug: Symptomatic treatment (paracetamol or best symptomatic treatment based on doctor recommendations)

INTERVENTIONS:
Drug: Colchicine plus symptomatic treatment (paracetamol) — Colchicine plus symptomatic treatment (paracetamol).
  Arms: Colchicine plus symptomatic treatment (paracetamol).
Drug: Symptomatic treatment (paracetamol or best symptomatic treatment based on doctor recommendations) — Symptomatic treatment (paracetamol or best symptomatic treatment based on doctor recommendations).
  Arms: Symptomatic treatment

SUMMARY:
This is a phase 3 clinical trial, randomized, single-center, opened, controlled, to evaluate efficacy and safety of early administration of colchicines in patients older than 60 years, with high risk of pulmonary complications due to coronavirus SARS-CoV2 (COVID-19). An approximately number of 954 subjects meeting all inclusion and none exclusion criteria will be randomized either to receive colchicines or symptomatic treatment with paracetamol during 21 days.

DETAILED DESCRIPTION:
The primary objective of the study is to determine whether short term course of colchicines reduces number of deaths due to COVID-19 and severe complications due to the virus in elderly patients with comorbidities.

The secondary objective is to determine the safety of colchicines in this patient population.

Approximately 954 subjects who meet all inclusion criteria and none exclusion criteria will be randomized either to receive colchicines or symptomatic treatment (2:1 allocation ratio) during 21 days. Follow-up assessments will occur every 48 hours and always at day 10, 21 and 61 following randomization for evaluation of the occurrence of any trial endpoints or other adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes who are at least 60 years old.
2. Diagnosis of COVID-19 infection in the last 72 hours and confirmed by PCR
3. Patient in outpatient follow-up (not hospitalized or under consideration) or institutionalized in senior centers/residences
4. The patient must possess at least two of the following high-risk criteria

   1. 60 years of age or older AND
   2. Any of the following: Diabetes mellitus, high blood pressure, known pulmonary disease (including asthma or chronic obstructive pulmonary disease), known heart failure, known coronary disease, bicytopenia, pancytopenia, or the existence of simultaneous neutrophilia and lymphopenia
5. The patient must be able and willing to comply with the requirements of this study protocol.

Exclusion Criteria:

1. Hospitalized patient or under immediate consideration of doing so
2. Patient taking colchicine for other indications
3. Patient with history of allergic reaction or sensitivity to colchicine
4. Patient with inflammatory bowel disease, gastric ulcer, chronic diarrhea or malabsorption
5. Patient with pre-existing progressive neuromuscular disease
6. Patient with kidney damage and estimated glomerular filtrate rate <30 ml/m at 1732
7. Patient undergoing chemotherapy for cancer, including haematological malignancies.
8. Patients being treated with CYP3A4 and/or glycoprotein inhibitor drugs
9. Immunosuppressive treatment
10. History of cirrhosis, chronic active hepatitis, severe chronic disease defined by GOT or GPT values exceeding 3 times the upper limit of normal.
11. If the investigator considers it, for any reason, to be an inadequate candidate.
12. Patient and/or legal representative will not have signed the informed consent form.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Number of participants who die due to COVID-19 infection | 21 days post-randomization
Number of participants who require hospitalization due to COVID-19 infection | 21 days post-randomization

OTHER OUTCOMES:
A confirmed diagnosis from COVID-19 infection (by positive PCR test) will be mandatory . | 48 hours
  not delayed more than 48 hours from initial symptoms

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Atención primaria (Área 2), Laredo, Cantabria
  - Gerencia de atención primaria (Área 3), Reinosa, Cantabria
  - Atencion primaria (AREA 1), Santander, Cantabria
  - Gerencia de atención primaria (área 4), Torrelavega, Cantabria

REFERENCES:
- [Derived] Estebanez EB, Alconero LL, Fernandez BJ, Marguello MG, Caro JCL, Vallejo JD, Sampedro MF, Cacho PM, Espiga CR, Saiz MMG. The effectiveness of early colchicine administration in patients over 60 years old with high risk of developing severe pulmonary complications associated with coronavirus pneumonia SARS-CoV-2 (COVID-19): study protocol for an investigator-driven randomized controlled clinical trial in primary health care-COLCHICOVID study. Trials. 2021 Sep 6;22(1):590. doi: 10.1186/s13063-021-05544-7. PMID 34488841